CLINICAL TRIAL: NCT03686267
Title: Evaluation of the Esthetic Outcome of Lithium Disilicate (e.Max) All Ceramic Crowns on Titanium Implant Abutments in the Esthetic Zone After Different Color Masking Approaches; a Randomized Clinical Trial
Brief Title: Evaluation of the Aesthetic Outcome of Lithium Disilicate (e.Max) All Ceramic Crowns on Titanium Implant Abutments in the Aesthetic Zone After Different Color Masking Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karim Ahmed Awadallah Osman, assistant lecturer- fixed prosthodontics department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CEBD-CU-2018-09-26
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Aesthetic Outcome of Crowns on Implants
Keywords: implants- titanium abutments- all ceramic crowns- lithium disilicate- color measurements- pink and white aesthetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: TRIPLE BLINDED
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention (I1) (Experimental): Lithium disilicate crowns over titanium abutments covered by a layer of opaque porcelain
  Interventions: Other: opaqued titanium abutments
- Intervention (I2) (Experimental): Lithium disilicate crowns over titanium abutments covered by lithium disilicate (high opacity) coping
  Interventions: Other: lithium disilicate coping (high opacity)
- Lithium disilicate crowns over uncovered titanium abutments (Active Comparator): Lithium disilicate crowns over uncovered titanium abutments directly without masking
  Interventions: Other: titanium abutment with no color masking

INTERVENTIONS:
Other: opaqued titanium abutments — masking metallic color of titanium abutments by opaque porcelain
  Arms: intervention (I1)
Other: lithium disilicate coping (high opacity) — masking metallic color of titanium abutments using lithium disilicate copings
  Other Names: E-max coping
  Arms: Intervention (I2)
Other: titanium abutment with no color masking — color masking methods are avoided in this arm
  Arms: Lithium disilicate crowns over uncovered titanium abutments

SUMMARY:
Implants have become the perfect solution for replacement of missing single teeth, partial or even complete edentulism.18 However, the dilemma of anterior implant-supported prosthesis is still not quite solved.19-21 Implant abutments are one of the esthetic influencers. And concerning the material, ready-made titanium abutments are considered the gold standard of all. Nevertheless, the esthetic properties remain doubtful. Lithium disilicate ceramics have been used as implant superstructures for many years now for their combined esthetic and biomechanical properties. The purpose of the present study is to evaluate the effect of using titanium implant abutment on the color of lithium disilicate crowns and the significance of masking the titanium abutments with opaque porcelain or using opaque lithium disilicate coping on the final esthetic outcome

DETAILED DESCRIPTION:
Clinical resemblance is one the of main factors that preclude the success of any restoration. The use of conventional titanium implant abutment and ceramic restoration succeeded to prevail until now. New ceramic and polymer derivatives have been introduced such as hybrid ceramics, PEEK and PEKK. However, the low mechanical properties and the ease of breakage still limited them to certain clinical situations. Hybrid fixture-abutment combinations such as hybrid abutments and hybrid crowns proved to be highly efficient in the literature. But the technique sensitivity and the urge of high clinical and laboratory skills are obstacles that must be taken into consideration. This is the reason that finding esthetic modification of the conventional techniques seems reasonable. Masking the color of the underlying abutment appears to be a simple and easily achievable solution for having a highly esthetic implant supported prosthesis.

The importance of peri-implant soft tissues, whether esthetically or biologically, has been emphasized in literature. (4) Furthermore, achieving the desired esthetic outcome depends on simultaneously matching the proper esthetic criteria of the tooth and its supporting structures. (5) Esthetic failures in implant dentistry can be categorized as pink-tissue failures and white-tissue failures. (6) Pink esthetics include color, texture and level of peri-implant tissues (7), while white esthetics include color, shape and characterization of crown. (3) The mode of fabrication also influences the performance of the materials, where the use of press technology facilitates the construction of implant supported crowns, offering precision of fit, durability and esthetic materials application. (11)

ELIGIBILITY:
Inclusion Criteria:

* 1. Above 18 years old 2. Literate, capable of reading and signing the informed consent document 3. Healthy, Free from or with controlled systemic disease 4. With acceptable oral health to support implant restorations 5. With good bone quality and quantity 6. Cooperative, accepting follow up and maintenance sessions 7. Having missing tooth in esthetic zone

Exclusion Criteria:

* 1. Under 18 years old 2. Illiterate, unable of comprehending or signing the informed consent document 3. Unhealthy with uncontrolled systemic disease (e.g. Diabetes or hypertension) 4. Pregnancy 5. With unfavorable oral state that might affect implant procedure and restoration 6. Uncooperative, not willing to return for follow up visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Pink esthetics and White esthetics | six months
  using numerical score (0-10) to evaluate the aesthetics of soft and hard dental tissues

SECONDARY OUTCOMES:
Color measurements | six months
  using Spectrophotometer to evaluate color in terms of CIE L* a* b* values

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided